CLINICAL TRIAL: NCT02515903
Title: Comparison Between Stereotactic Aspiration and Intra-endoscopic Surgery to Treat Intracerebral Hemorrhage
Acronym: EndoSurofICH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFYY-NSD-001
Record Dates: First submitted 2015-07-22; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Intracerebral Hemorrhage; Surgery
Keywords: Endoscopy; Intracerebral hemorrhage; surgery; stereotactic aspiration; Key-hole approach; Intracerebral hemorrhage surgical treatment; Transparent endoscopic sheath; Agitation-aspiration device
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-endoscopy (Experimental): This intervention arm will receive intra-endoscopic evacuation surgery for ICH.
  Interventions: Procedure: Intra-endoscopic surgery
- Stereotactic Aspiration (Placebo Comparator): This arm will receive stereotactic aspiration surgery for ICH evacuation.
  Interventions: Procedure: Placebo:stereotactic aspiration surgery

INTERVENTIONS:
Procedure: Intra-endoscopic surgery — Intra-endoscopic surgery for evacuation of ICH
  Arms: Intra-endoscopy
Procedure: Placebo:stereotactic aspiration surgery — Placebo:stereotactic aspiration surgery for evacuation of ICH
  Arms: Stereotactic Aspiration

SUMMARY:
Views for surgery method selection of intracerebral hemorrhage are still controversial. Since the application of neuroendoscopic technique in intraventricular hemorrhage was confirmed effective and safe, some investigators have attempted to use endoscopic strategies to evacuate intracerebral hematomas. Some significant advances have also been reported in endoscopic hematoma evacuation when compared to conventional craniotomy. However, it is still crucial to implement a prospective and controlled study to evaluate the efficiency and safety of endoscopic technique in the treatment of intracerebral hemorrhage. In this study, the investigators will exclusively select some patients with intracerebral hemorrhage in the basal ganglia region. This study will compare the efficacy and safety of endoscopic surgery versus stereotactic aspiration on neurologic outcomes for patients with intracerebral hemorrhage.

DETAILED DESCRIPTION:
Although the incidence and mortality of spontaneous intracerebral hemorrhage (ICH) have been decreased with the improved management of high blood pressure, ICH may induce serious disability for the patients and continue to be a major socioeconomic problem. The evacuation of ICH using open craniotomy or computer tomography (CT)-guided stereotaxy may improve the survival rate of these patients but failed to prove efficacy in improving patients' functional outcome despite numerous efforts. Endoscopy-guided evacuation of ICH provides a less invasive and quicker surgical decompression, which may potentially improve the functional outcome for patients. In previous studies, endoscope-guided evacuation of ICH is often referred to as that an endoscope only provides an illuminating system while the operating channel is independent from the endoscope (endoscopy-controlled microneurosurgery or endoscopy-assisted microneurosurgery). In recent years, authors have been committed to explore the procedure of intra-endoscopy-guided evacuation of ICH, which means that the illuminating channel, the irrigation-aspiration channel and the working channel are all located in the endoscope. This kind of procedure can be called as real endoscopic neurosurgery (EN), which may potentially decrease the operative concomitant injuries at the most extent. However, the inherent drawbacks of intra-endoscopic procedures, including the limited visualization of the surgical field and the difficult maintenance of patency of the aspiration wand, can offset the advantages in some instances. The authors exclusively invented a special endoscopic transparent sheath for guiding hematoma puncture and an agitation-aspiration system (AAS) for keeping patency of the aspiration wand. Detailed procedures of their application will be implemented and verified in a series of patients with intracerebral hemorrhage. Meanwhile, the mortality rate, complications and other outcome parameters between this procedure and CT-guided procedures will be compared.

ELIGIBILITY:
Inclusion Criteria:

* primary basal ganglion region intracerebral hemorrhage
* older than 18 years
* admitted within 6 h after onset of ICH

Exclusion Criteria:

* other type of ICH than acute primary intracerebral hemorrhage
* patients who need neurosurgery
* life expectancy less than 3 months due to comorbid disorders
* confirmed malignant disease (cancer)
* confirmed acute myocardial infarction
* hepatitis and/liver cirrhosis
* renal failure
* infectious disease (HIV, endocarditis etc.)
* current or previous hematologic disease
* women of childbearing age if pregnant
* participation in another study within the preceding 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 90-day
  all-cause motality rate within 90 days after the surgery

SECONDARY OUTCOMES:
operative time | 24 h
  the period from skin incision to wound suture
days of ICU stay | 14 day
  the period between the end of the surgery to leaving the ICU
remnant blood in the hematoma after surgery | 12 hour
  this parameter will be monitored by CT scan immediately after the surgery
Glasgow coma score | 28 day
  the GCS will be evaluated by a senior doctor 28 days after the surgery
Glasgow outcome score | 90-day
  the GCS will be evaluated by a senior doctor 28 days after the surgery
In-hospital cost | 28 day
  all medical cost during the in-hospital period
rehemorrhage rate | 3 day
  Rehemorrhage almost occurs within 3 days after the surger. So cranial CT scan will be performed routinely 3 days later after surgery to evaluate the rehemorrhage rate
intracranial infection | 14 day
  If the patient underwent a period of fever, cerebral fluid will be withdrawn by means of lumbar puncture and tested to verify whether the intracranial infection occurs

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Du B, Xu J, Hu J, Zhong X, Liang J, Lei P, Wang H, Li W, Peng Y, Shan A, Zhang Y. A Clinical Study of the Intra-Neuroendoscopic Technique for the Treatment of Subacute-Chronic and Chronic Septal Subdural Hematoma. Front Neurol. 2020 Jan 17;10:1408. doi: 10.3389/fneur.2019.01408. eCollection 2019. PMID 32010057
- [Derived] Zhang Y, Shan AJ, Peng YP, Lei P, Xu J, Zhong X, Du B. The intra-neuroendoscopic technique (INET): a modified minimally invasive technique for evacuation of brain parenchyma hematomas. World J Emerg Surg. 2019 May 6;14:21. doi: 10.1186/s13017-019-0239-0. eCollection 2019. PMID 31080494
- [Derived] Du B, Shan AJ, Zhang YJ, Wang J, Peng KW, Zhong XL, Peng YP. The intra-neuroendoscopic technique: A new method for rapid removal of acute severe intraventricular hematoma. Neural Regen Res. 2018 Jun;13(6):999-1006. doi: 10.4103/1673-5374.233442. PMID 29926826